CLINICAL TRIAL: NCT06539442
Title: Prospective Clinical Study to Assess the Safety and Efficacy of Versius, in Urological Procedures in Paediatrics
Brief Title: Versius Paediatrics Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMR Surgical Ltd (Industry)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-00533
Record Dates: First submitted 2024-07-24; First posted 2024-08-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Robotic Surgical Procedures in Pediatric Urology
Keywords: Pediatric; Paediatric; Versius; Urology; Robotic assisted surgery; minimal access surgery; minimally invasive surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Versius Surgical System (Experimental)
  Interventions: Device: Versius Surgical System

INTERVENTIONS:
Device: Versius Surgical System — Urological minimal access surgery performed with Versius Surgical System

SUMMARY:
This is prospective, multi-phase, single arm, multi-centre, multi-surgeon feasibility clinical trial to provide proof of concept and clinical evidence regarding the safety and efficacy of Versius (robotic surgery medical device) in Urological Procedures in Paediatric population. In alignment with IDEAL (Idea, Development, Exploration, Assessment, Long-term study) Framework, this study will consist of 3 main phases to ensure proper procedure development while ensuring patients safety. Feasibility and safety will be assessed on an ongoing basis, and specifically after completion of the first 3 procedures, at a single site (Southampton/Lead), each conducted one week apart to allow the identification of unanticipated risks/adverse events. Once deemed safe, based on the results of the 3 cases enrolled in Phase I, 7 further cases would be completed, at the same site. Once the procedure is deemed safe according to safety data collected, the recruitment will proceed to full trial patient accrual, 140 additional cases from the 3 participating study sites.The study patient population is children and adolescents under the age of 18, which will be provided clinical care and follow-ups per standard of care and hospital's policy.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, (<18 years old) for whom an appropriate legal representative provides written consent for participation
* Patient and disease factors deemed suitable for minimal access urological procedure
* Multidisciplinary team (MDT) decision to treat with surgery
* Patients under the care of the paediatric urology team in one of the participating centres

Exclusion Criteria:

* Patients ≥ 18 years old
* Appropriate legal representative unwilling to provide written consent
* Medical contraindication for general anaesthesia
* Medical contraindication for laparoscopic procedure
* Active pregnancy (in post-pubertal female patients)
* Morbid obesity (BMI ≥ 40 kg/m2)
* Patient participation in an interventional clinical study, that could impact primary objectives results
* Prior pelvic /abdominal radiotherapy treatment
* Subjects with other clinically significant unstable medical disorder, life-threatening disease, or anything else in the opinion of the Investigator which would contra-indicate a surgical procedure

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event rate | Up to 3 months post operation
  Incidence of adverse events

SECONDARY OUTCOMES:
Procedure completion | Day of operation
  Rate of successful completion of procedures without unplanned conversion to other laparoscopic or open surgery
Serious Adverse Event Rate | Up to 3 months post-operation
  Incidence of serious adverse events
Ultrasound grading | 3 months post stent removal
  Ultrasound hydronephrosis grading results
MAG3 Renogram | 3 months post stent removal
  MAG3 Renogram results
Operative time | Day of operation
  Surgery duration from skin incision to skin closure in minutes
Blood loss | Day of operation
  Estimated blood loss in mL
Post operative analgesic treatment | Immediately after surgery
  Pain medication prescribed post-operatively
Length of stay | Up to 3 months post operation, average 1 day
  Hospital stay from end of surgery to discharge in days
Reoperation | 24 hours post operation
  Reoperation within 24 hours of surgery
Unplanned readmission | Up to 3 months post operation
  Unplanned hospital readmissions
Device deficiencies and user errors | Day of operation
  Device deficiencies and user errors that occur during surgery
Ultrasound grading | 12 months post operation
  Ultrasound hydronephrosis grading results

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Brownlee, MD, Principal Investigator — Department of Paediatric Urology Southampton Children's Hospital; David Keene, MD, Principal Investigator — Department of Paediatric Urology Royal Manchester Children's Hospital; Pankaj Mishra, MD, Principal Investigator — Department of Paediatric Urology, Evelina London Children's Hospital
Locations (3):
- United Kingdom (3):
  - Department of Paediatric Urology, Evelina London Children's Hospital, London
  - Department of Paediatric Urology Royal Manchester Children's Hospital, Manchester
  - Department of Paediatric Urology Southampton Children's Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No